CLINICAL TRIAL: NCT02198846
Title: A Study to Compare the Efficacy and Safety of Insulin Pump Treatment in Patients With Uncontrolled Type 2 Diabetes Mellitus
Brief Title: A Study to Compare Insulin Pump With Conventional Treatment in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Soo Bong Choi, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU_PUMP1
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin pump (Experimental): insulin pump
  Interventions: Device: insulin pump
- conventional treatment (Active Comparator): intensification of conventional treatment
  Interventions: Drug: conventional treatment

INTERVENTIONS:
Device: insulin pump — stop any antihyperglycemic medication and convert to insulin pump
  Arms: Insulin pump
Drug: conventional treatment — intensification of conventional treatment by adding oral antihyperglycemic agents or subcutaneous insulin (once / twice/ multiple injection)
  Arms: conventional treatment

SUMMARY:
Insulin deficiency resulted from progressive beta cell failure and insulin resistance in type 2 diabetes requires exogenous insulin therapy, escaping from oral antihyperglycemic agents. Previous data have been suggested that continuous subcutaneous insulin infusion (CSII) does not only have efficacy in glucose control but also restore beta cell failure.

The investigators plan to compare the efficacy/safety and beta cell function between insulin pump treatment and the intensification of conventional treatment in patients with uncontrolled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age: 18 ~ 85 yrs
* HbA1c: > 7.5%
* no change of anti-diabetic medication within 3 months

Exclusion Criteria:

* systemic corticosteroid administered within previous 6 months
* pregnancy
* severe liver or renal disease, heart failure
* History of cancer within 5 years
* Thyroid disease
* Anti-obesity drugs or slimming products within previous 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
change of HbA1c | 24 weeks

SECONDARY OUTCOMES:
changes of body weight | 24 weeks
frequency of hypoglycemia | 24 weeks
  severe hypoglycemia : glucose <40 mg/dl mild hypoglycemia : glucose 40 - 70 mg/dl
change of beta cell function | 24 weeks
  insulin secretion-sensitivity index-2
  = insulinogenic index x Matsuda index
Percent of patients who reach target goal of HbA1c (<7.0%) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo Bong Choi, MD.PhD, Principal Investigator — Konkuk University
Locations (1):
- Konkuk University Chungju Hospital, Chungju, South Korea